CLINICAL TRIAL: NCT04953052
Title: A Randomized, Double-blind, Multicentre 2-arm, Parallel-group, Placebo-controlled Study to Investigate the Efficacy and Safety of Intravenous Imatinib Mesylate in Reducing the Severity of Hypoxemic Respiratory Failure in Patients With Critical COVID-19 Receiving Standard of Care.
Brief Title: A Randomized Study to Investigate the Effect of Intravenous Imatinib on the Amount of Oxygen in the Lungs and Blood of Adults With COVID-19 Needing Mechanical Ventilation and Supportive Care.
Acronym: IMPRESS COVID
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Number of moderate to severe ARDS patients hospitalised due to COVID19 diminishingly small. Not expected to recruit required minimum number of patients.
Sponsor: Exvastat Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EX003; 959310 (Other Grant/Funding Number: European Innovation Council Accelerator Grant)
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19 Acute Respiratory Distress Syndrome; Covid19; ARDS; Pulmonary Oedema
Keywords: Acute Respiratory Distress Syndrome; ARDS; Covid-19; Imatinib; Oxygen Saturation Index; OSI; Endothelial Dysfunction; Pulmonary Oedema; Protein Kinase Inhibitor
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Pulmonary Edema | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Imatinib Mesylate (Experimental): Intravenous Imatinib Mesylate solution- 200mg as an 8mg/ml solution, administered twice daily (400mg total daily dose). Each dose administered in a 25ml solution over a two-hour infusion period.
  Interventions: Drug: Imatinib Mesylate
- Intravenous Placebo (Placebo Comparator): Intravenous Placebo matched solution- administered 25ml solution, twice daily over a two-hour infusion period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imatinib Mesylate — An isotonic sterile solution of imatinib.
  Other Names: Impentri
  Arms: Intravenous Imatinib Mesylate
Drug: Placebo — An isotonic sterile solution
  Arms: Intravenous Placebo

SUMMARY:
The COVID-19 pandemic has led to an increase in the number of patients admitted to intensive care units (ICU) with acute respiratory distress syndrome (ARDS). ARDS is a severe, life-threatening medical condition characterised by inflammation and fluid in the lungs. There is no proven therapy to reduce fluid leak, also known as pulmonary oedema, in ARDS. However, recent studies have discovered that imatinib prevents fluid leak in the lungs in inflammatory conditions, while leaving the immune response intact.

Adding imatinib into the standard care package may, therefore, decrease mortality and reduce the duration of mechanical ventilation compared with standard care alone, in critically-ill patients with COVID-19.

To help determine the impact of imatinib in these patients we present a randomised, double-blind, multi-centre, 2-arm, parallel-group, placebo-controlled clinical study of intravenous imatinib in 84 mechanically-ventilated, adult subjects with COVID-19-related ARDS.

Study participants (patients who have consented into the study) will receive the study drug (imatinib or placebo) twice daily for a period of 10 days. The effect of the intervention will be tested by measuring the change from baseline in the Oxygen Saturation Index (OSI) at day 10. OSI is a non-invasive means of measuring oxygenation and is an independent predictor of mortality in patients with ARDS, serving thus as a relevant endpoint from which to assess the efficacy of imatinib.

Other measurements will include regular blood tests as part of safety assessments.

Time on ventilation and morbidity and mortality will be recorded as secondary outcome measures.

Blood tests will also allow the investigation of the pharmacokinetic properties of imatinib, as well as biomarkers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years
2. Women of childbearing potential must have a negative serum pregnancy test to confirm eligibility
3. Provision of signed written informed consent from the patient or patient's legally acceptable representative
4. SARS-CoV-2 infection confirmed by RT-PCR laboratory test (which may include results from a test that was performed prior to hospital admission if, in the opinion of the Investigator, it is relevant to ongoing COVID-19)
5. Meet Berlin definition for moderate - severe ARDS

   1. Bilateral opacities - not fully explained by effusions, lobar/lung collapse, or nodules
   2. Respiratory failure not fully explained by cardiac failure or fluid overload.
   3. PaO2/FIO2 ≤200 mmHg with PEEP ≥5 cmH2O
6. Patient requires intubation or is currently intubated and has been for ≤48 hours

Exclusion Criteria:

1. Persistent septic shock (>24 hours) with a Mean Arterial Pressure (MAP) ≤65 mm Hg and serum lactate level >4 mmol/L (36 mg/dL) despite adequate volume resuscitation and vasopressor use (norepinephrine >0.2 μg/kg/min) for >6 hours
2. Major trauma in the past 5 days
3. Presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the last year
4. Pre-existing severe cardiopulmonary disease including, but not limited to, interstitial lung disease; severe COPD (GOLD Stage IV or FEV1<30% predicted); heart failure (estimated left ventricular ejection fraction < 40%); or a chronic lung condition requiring home oxygen treatment
5. An underlying clinical condition that, in the opinion of the Investigator, would make it very unlikely for the patient to be successfully weaned from ventilation due to severe underlying diseases (e.g., severe malnutrition, severe neurological disease)
6. Patients considered inappropriate for critical care (e.g., being considered for palliative care)
7. Currently receiving extracorporeal membrane oxygenation (ECMO)
8. Severe chronic liver disease with Child-Pugh score >12 (Appendix 1)
9. White blood count <2.5 x 109/L; Hemoglobin <4.0 mmol/L (6.5g/dL); Platelets <50 x 109/L
10. ALT or AST >10x upper limit of normal (ULN) or bilirubin >3x ULN
11. Women who are pregnant or breast-feeding
12. Use of drugs with strong CYP3A4 induction potential, such as carbamazepine, efavirenz, enzalutamide, phenobarbital, phenytoin, hypericum, mitotane, nevirapine, primidone, rifabutin and rifampicin
13. Inability of the ICU staff to initiate administration of study treatment within 48 hours of intubation
14. Enrolled in a concomitant clinical trial of an investigational medicinal product
15. In the opinion of the investigator, progression to death is highly probable, irrespective of the provision of treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-14 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Oxygen Saturation Index (OSI) at Day 10 | From Baseline to Day 10
  Oxygen saturation is a calculation derived from [mean airway pressure × FiO2 × 100] / SpO2.

SECONDARY OUTCOMES:
Change from Baseline in Oxygen Saturation Index (OSI) at Day 3 and Day 5 | From Baseline to Day 3 and from baseline to Day 5
  Oxygen saturation measured by pulse oximetry
Mortality rate at Day 29 and Day 60 | Day 29 and Day 60
  Mortality at Day 29 and Day 60
Change from baseline in WHO 9-point ordinal scale for clinical improvement to Day 10 and Day 29 | The WHO ordinal scale will be recorded Days 1-10 and Day 29
  The WHO Ordinal Scale for Clinical Improvement (0 to 8, where a higher value indicates worse outcome).
  It measures illness severity over time using the following categories: Uninfected, Ambulatory (no limitation of activities), Ambulatory (limitation of activities), Hospitalized (no O2 therapy), Hospitalized (O2 by nasal prongs or mask), Hospitalized (O2 by NIV or HFNO), Hospitalized (intubation and invasive mechanical ventilation), Hospitalized (ventilation and additional organ support [vasopressors, CVVH, ECMO]), Death.
Duration of mechanical ventilation (Days) to Day 29 and Day 60 | To Day 29 and to Day 60
  Number of days requiring to be on mechanical ventilation
Duration of stay in ICU (Days) to Day 29 and Day 60 | To Day 29 and to Day 60
  Number of days within the ICU
Time to first successful extubation (Hours) to Day 29 | To Day 29
  Number of hours to extubation (removal of the endotracheal tube)
Number of days free of mechanical ventilation and survival (VFDsurv) at Day 29 and Day 60 | At Day 29 and Day 60
  Amongst survivors, the number of days free from mechanical ventilation

OTHER OUTCOMES:
Safety- Type, frequency, severity, and relationship to study treatment of any AEs, SAEs or AEs leading to discontinuation of study treatment from Day 1 to Day 29 (final follow up visit) | Day 1 to Day 29
  Safety adverse events and serious adverse event collection
Incidence of related Treatment-Emergent Adverse Events- Tolerability | Day 1 to Day 29
  Tolerability
Pharmacokinetic- Imatinib plasma concentration | 4 samples collected Day 1, and single samples collected Days 3 and 5
  Imatinib plasma concentration- Multivariate hierarchical analysis will be performed on various factors (age, sex, weight, height,appha-1-acid glycoprotein, haemoglobin, ALAT, CRP, eGFR, albumin, smoking, and concomitant drugs) to explore sources of variability in patient outcome. Significant predictors will be used as covariates to improve the performance of the PK model.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Burgess, MD, Study Director — Exvastat Ltd.
Locations (8):
- India (8):
  - Sir Sayajirao General Hospital (SSG Hospital), Medical College Baroda, Jail Road Indira Avenue)Anandpura, Vadodara, Gujarat
  - St George's Hospital, P D Mello Road, Fort Road, CST Terminal,, Mumbai, Maharashtra
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - PCMC PGI Yashwantrao Chavan Memorial Hospital, Nagar, Pune
  - NRS Medical College and Hospital, Kolkata, West Bengal
  - Father Muller Hospital and Medical College, Mangalore
  - JSS Hospital, Mysuru
  - Indira Gandhi Government Medical College and Hospital, Nagpur

IPD SHARING:
Plan to Share IPD: Undecided